CLINICAL TRIAL: NCT04718233
Title: Effect of Sildenafil Citrate on Mid Luteal Phase Uterine Artery Blood Flow in Patients With Recurrent Pregnancy Loss Due to Impaired Uterine Artery Blood Flow
Brief Title: Effect of Sildenafil Citrate on Mid Luteal Phase Uterine Artery Blood Flow in Patients With Recurrent Pregnancy Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Abass, lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: sildenafilcitrate89
Record Dates: First submitted 2021-01-16; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Recurrent Pregnancy Loss
MeSH Terms: interventions — Sildenafil Citrate; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sildenafil citrate (Experimental): Sildenafil citrate at a dose of 25mg will be administered orally in patients with recurrent pregnancy loss and the blood flow indices will be measured initially and after 3 hours.
  Interventions: Drug: Sildenafil 25Mg Tablet
- placebo (Placebo Comparator): placebo will be administered orally in patients with recurrent pregnancy loss and the blood flow indices will be measured initially and after 3 hours.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Sildenafil 25Mg Tablet — Sildenafil citrate at a dose of 25mg will be administered orally in patients with recurrent pregnancy loss
  Arms: sildenafil citrate
Drug: Placebo Oral Tablet — placebo will be administered orally in patients with recurrent pregnancy loss
  Arms: placebo

SUMMARY:
Patients with recurrent pregnancy loss are known to have decreased uterine artery blood flow. Nitric oxide plays a major role in increasing uterine blood flow during the luteal phase. This study is done to evaluate the effects of sildenafil on blood flow indices in the patients with recurrent pregnancy loss due to impaired uterine artery blood flow.

DETAILED DESCRIPTION:
Study Setting: The study will be conducted in recurrent pregnancy loss outpatient clinic at Ain shams university maternity hospital.

Study Population: Patients with unexplained recurrent miscarriage attending Ain shams university maternity hospital's outpatient clinic. This study will be conducted on 80 women distributed into 2 groups each is 40 women in fertile age with history of two or more recurrent spontaneous abortions and decreased uterine artery blood flow(PI>2.02(Mansour et al., 2018). First group will be placebo controlled and the second group will be given sildenafil citrate.

Women will be asked to attend during the 21-23 day of the cycle and will be subjected to: History taking and Full clinical examination.

Clinical examination will be done including general, abdominal and pelvic examination.

General examination: including general appearance, weight, height and vital signs Abdominal examination: to assure freedom of any organic clinically detectable pathologic lesions.

Pelvic examination: included inspection of the external genitalia, speculum examination of the vagina to rule out infection, and bimanual assessment of uterine size and position as well as exclusion of adnexal masses.

Laboratory investigations:

Routine investigations including: CBC, fasting and postprandial blood sugar, urine analysis, kidney function and liver function will be done.

The endocrine evaluation consisted in measuring thyroid-stimulating hormone, free thyroxin, and progesterone levels on day 21 of the menstrual cycle.

Sonography:

Sonography will be performed using Samsung H60 with convex probe (multi-frequency AD 2~ 8 MHz) to perform trans-vaginal examination. Examination will be performed in the second phase of the menstrual cycle, at mid-luteal day.

Pulsed wave Doppler will be used to obtain clear, consistent, flow velocity wave forms of both uterine arteries. Pulsatility index (PI) will be measured bilaterally. The PI reported will be the arithmetic mean for the last three cardiac cycles.

(Goswamy and Steptoe, 1988) classification will be used to determine the wave types. According to this classification, the FVW of the circumflex artery can be of 3 types : Type A when the diastolic component is present but not continuous with the systole, and ends before the next cardiac cycle.

Type B when a diastole is present and continues with the systole, but ends before the next cardiac cycle.

Type C when a diastole is present and continues with the systole and into the next cardiac cycle.

The majority of research has centered on an elevation in the RI or PI to detect the presence of increased uterine artery blood flow resistance in non- pregnant states. Criteria for an abnormal uterine artery Pulsatility index (PI) cutoff (PI> 2.02) and abnormal sub-endometrial blood flow Resistant Index (RI) (RI>0.6) (Mansour et al., 2018).

Steps and methods:

The participants will be two groups of 80 patients with history of recurrent pregnancy loss, each is 40.

All patients will be scanned transvaginally with transvaginal Doppler sonography 6 to 8 days after ovulation to measure the pulsatility index (PI), resistance index (RI) and systolic to diastolic ratio (S/D) of the right and left main uterine arteries and sub-endometrial blood flow resistance index (RI). Sildenafil citrate at a dose of 25mg or placebo will be administered orally in patients with recurrent pregnancy loss and the blood flow indices will be measured after 3 hours. The student test will be used for analysis of the results, P< 0.05 will be considered significant.

With 95% confidence interval. P values ≥5% considered to be significant.

ELIGIBILITY:
Inclusion Criteria:

1. History of 2 or more unexplained recurrent miscarriage.
2. Child bearing period (18-35 years old).
3. Non pregnant state.
4. Regular menstrual cycles for the previous three months before the study.
5. No hormonal contraception or intrauterine device.
6. impaired uterine artery blood flow (PI >2.02) (Mansour et al., 2018).

Exclusion Criteria:

* 1-Having any possible causes of abortion: anatomical, genetic, endocrinological, infectious, or immunological.

  2- Autoimmune disorders which may affect blood vessels and their blood flow (systemic lupus).

  3- Systemic disease that might affect the hemodynamic indices (e.g. thrombocytopenia, thyrotoxicosis … etc.).

  4- Diagnosed or treated thrombophilia. 5- Any vascular disease (e.g. coronary artery disease). 6- History of oophorectomy. 7- History of consanguinity. 8- Family history of chromosomal abnormalities (e.g. trisomy 21, trisomy 13… etc.).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
uterine artery blood flow indices | 3 hours
  uterine artery PI, RI

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university maternity hospital, Cairo, Egypt